CLINICAL TRIAL: NCT06776887
Title: Virtual Reality-based Exercises on Postural Stability, Depressive Symptoms and Anxiety in Patients with Lower Extremity Burn: a Randomized Controlled Study
Brief Title: Virtual Reality-based Exercises on Postural Stability, Depressive Symptoms and Anxiety in Patients with Lower Extremity Burn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Abd el fattah Ali, Assistant Professor of physical therapy for surgery, Faculty of physical therapy-cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005525
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Patients with Lower Extremity Burn; Postural Stability, Depressive Symptoms and Anxiety in Patients with Lower Extremity Burn
Keywords: Virtual reality-based exercises -Postural stability, depressive symptoms- anxiety - lower extremity burn
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Forty patients of both sexes with healed LL burn will be divided into two groups:
  The Wii Fit group will receive the Wii Fit program for 30 minutes in addition to SPTP for 60 minutes, whereas. The intervention was 3 sessions a week for 12 weeks.
  The control group will receive standard physical therapy program (SPTP) only 3 sessions a week for 12 weeks
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A(Wii fit group) (Experimental): The Wii Fit group will receive the Wii Fit program for 30 minutes in addition to SPTP for 60 minutes, whereas. The intervention was 3 sessions a week for 12 weeks.
  Interventions: Device: The Wii Fit group will receive the Wii Fit program for 30 minutes in addition to SPTP for 60 minutes, whereas. The intervention was 3 sessions a week for 12 weeks
- group B(control group) (Active Comparator): The control group will receive standard physical therapy program (SPTP) only 3 sessions a week for 12 weeks .
  Interventions: Device: The Wii Fit group will receive the Wii Fit program for 30 minutes in addition to SPTP for 60 minutes, whereas. The intervention was 3 sessions a week for 12 weeks

INTERVENTIONS:
Device: The Wii Fit group will receive the Wii Fit program for 30 minutes in addition to SPTP for 60 minutes, whereas. The intervention was 3 sessions a week for 12 weeks — The Wii Fit group will receive the Wii Fit program for 30 minutes in addition to SPTP for 60 minutes, whereas. The intervention was 3 sessions a week for 12 weeks.
  The control group will receive standard physical therapy program (SPTP) only 3 sessions a week for 12 weeks .

SUMMARY:
A burn can be a life-threatening and traumatic event associated with severe pain and long-term health problems. Psychological difficulties are often reported after a burn, and symptoms of depression are one of the most common [1,2]. Physiological and state anxiety increased as a result of increased postural threat whereas ratings of perceived stability and balance efficacy were reduced as a function of increased postural threat. Efforts to diagnose balance disorders based on balance performance may be confounded by the influence of psychological factors. In a systematic review of the prevalence of depression after a burn, 4%-10% met the criteria for major depression within a year after the burn, and the rate of clinically relevant depressive symptoms measured by self-reporting was 4%-26% [3]. In addition, depressive symptoms after a burn have been associated with deterioration in long-term physical functioning and health-related quality of life (HRQoL) [[4], [5], [6]].

For patients with burns, studies have reported symptoms of anxiety in hospital [7,8], but Williams and Griffiths [9] reported that one third of a sample of 23 survivors of burns were still having appreciable psychological difficulties one year after the burn. Anxiety was the most common, followed by post-traumatic stress syndrome and depression Many treatments are available to treat anxiety and depression disorders, including medication, exercise, meditation, and cognitive behavioral therapy. In many cases, these treatments can be tailored to a client to help reduce symptomology of anxiety and/or depression. To date, the application of emerging technology in health promotion has generated substantial public interest. Among the emerging technologies that may potentially aid in the treatment of anxiety and depression, virtual reality (VR) is arguably the most exciting and technologically-advanced. VR is a digital technology that artificially creates sensory experiences-including visual, auditory, touch, and scent stimuli-while allowing the user to manipulate objects within the virtual environment created [3].

DETAILED DESCRIPTION:
A burn can be a life-threatening and traumatic event associated with severe pain and long-term health problems. Psychological difficulties are often reported after a burn, and symptoms of depression are one of the most common [1,2]. Physiological and state anxiety increased as a result of increased postural threat whereas ratings of perceived stability and balance efficacy were reduced as a function of increased postural threat. Efforts to diagnose balance disorders based on balance performance may be confounded by the influence of psychological factors. In a systematic review of the prevalence of depression after a burn, 4%-10% met the criteria for major depression within a year after the burn, and the rate of clinically relevant depressive symptoms measured by self-reporting was 4%-26% [3]. In addition, depressive symptoms after a burn have been associated with deterioration in long-term physical functioning and health-related quality of life (HRQoL) [[4], [5], [6]].

For patients with burns, studies have reported symptoms of anxiety in hospital [7,8], but Williams and Griffiths [9] reported that one third of a sample of 23 survivors of burns were still having appreciable psychological difficulties one year after the burn. Anxiety was the most common, followed by post-traumatic stress syndrome and depression Many treatments are available to treat anxiety and depression disorders, including medication, exercise, meditation, and cognitive behavioral therapy. In many cases, these treatments can be tailored to a client to help reduce symptomology of anxiety and/or depression. To date, the application of emerging technology in health promotion has generated substantial public interest. Among the emerging technologies that may potentially aid in the treatment of anxiety and depression, virtual reality (VR) is arguably the most exciting and technologically-advanced. VR is a digital technology that artificially creates sensory experiences-including visual, auditory, touch, and scent stimuli-while allowing the user to manipulate objects within the virtual environment created [3].

to our knowledge there is lack of studies assessing the effect of virtual reality based exercises on balance, depressive symptoms and anxiety in adult patients with lower extremity burn so this study is designed to assess the effect of virtual reality based exercises on balance, depressive symptoms and anxiety in adult patients with lower extremity burn

ELIGIBILITY:
Inclusion Criteria:

* age of the patient will be ranged from 35 to 55 years; 2) weight range 60-85 kg, height 155-170 cm; 3) total burned surface area (TBSA) was more than 40% measured by the rule of nines; 4) the burn cause was thermal; 5) burn depth, partial-thickness burn injury; 6) at least 3 months after burn injuries; 7) and with low physical activity level.

Exclusion Criteria:

* Patients will be excluded if they had 1) inhalation injury; 2) leg amputation; 3) any limitation in LL range of motion; 4) auditory or visual problems; 5) congenital musculoskeletal deformities, especially in the foot; 6) psychiatric disorders; 7) paralysis; or 8) cardiac abnormalities or cardiac pacemakers.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Biodex Balance System | 12 weeks
  Biodex Medical Systems, Shirley, NY) which consists of a movable balance platform that provides 20° surface tilt through 360° range of motion. The platform interfaces with computer software that enables the device to serve as an objective assessment of balance. All measurements were performed at level eight of stability, and the test duration was set at 20 seconds for three successive trials

SECONDARY OUTCOMES:
The Beck Depression Inventory-II (BDI-II) | 12 weeks
  has become one of the most widely used measures to assess depressive symptoms and their severity in adolescents and adults [9]. The BDI-II [5] is a 21-item self-report measure that taps major depression symptoms according to diagnostic criteria listed in the Diagnostic and Statistical Manual for Mental Disorders [10]. Items are summed to create a total score, with higher scores indicating higher levels of depression. It is worth noting that the BDI-II is not only extensively applied for research purposes but also in clinical practice, being the third test most used among Spanish professionals [11].
Anxiety was measured by the Dutch edition of the state version of the Spielberger State-Trait Anxiety Inventory (STAI). | 12 weeks
  This instrument is a 20-item measure of general anxiety and tension reflecting responses to situational factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study results
Supporting Information: Study Protocol